CLINICAL TRIAL: NCT04070014
Title: Relationship Between Heme Oxygenase 1 Enzyme Level and SYNTAX Score in Patients With Stable Coronary Artery Disease
Brief Title: Relationship Between Heme Oxygenase 1 Enzyme Level and Coronary SYNTAX Score
Status: Completed | Type: Observational
Sponsor: Yeditepe University Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Aytek Simsek, Assistant Professor, Yeditepe University Hospital
Other Study IDs: YeditepUH
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Coronary Artery Disease; Oxidative Stress
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum obtained from peripheral blood will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of this study is to investigate the relationship between heme oxygenase-1 enzyme level and angiographically determined SYNTAX score in patients with suspected stable coronary artery disease. Consecutive patients who are deemed to undergo coronary angiography due to high pre test probability or evidence of cardiac ischemia in imaging studies will be included in the study. Patients with coronary artery bypass surgery history and severe comorbid illnesses such as active malignancy, chronic obstructive lung disease, stage 3-5 chronic renal failure will be excluded. Serum heme oxygenase levels will be measured by ELISA method and SYNTAX score will be calculated from coronary angiography.

DETAILED DESCRIPTION:
Heme oxygenase-1(HO-1) is an enzyme found throughout the body with highest concentrations in tissues of reticuloendothelial system. It degrades heme to biliverdin and produces ferrous iron and carbon monoxide. It is an inducible anti oxidant enzyme production of which increases during high levels of oxidative stress. Synthesis of HO-1 is regulated mainly on transcriptional level.

Coronary artery disease is characterized by high oxidative stress levels. Initiation of atherosclerosis as well as progression and vulnerable plaque formation are shown to be linked to oxidation-anti oxidation imbalance.

Several studies showed a correlation between heme oxygenase-1 level, activity and coronary artery disease. Measuring heme oxygenase-1 activity from peripheral blood samples is technically challenging. Bilirubin levels are used as a marker of heme oxygenase activity and are showed to be related to coronary artery disease. As previously mentioned HO-1 is an inducible enzyme so the increased levels reveal a high oxidative stress situation. High levels of serum HO-1 are found also in other clinical settings such as interstitial pneumonia, malignancies, acute kidney injury.

Burden of coronary artery disease is highly correlated with adverse prognosis in patients with stable coronary artery disease and acute coronary syndrome. SYNTAX score is a well established tool to determine the extent of coronary artery disease. Severity and location of coronary stenoses as well as calcification and morphology are considered in SYNTAX score. Clinical SYNTAX score also incorporates clinical characteristics of patients including age, creatinine clearance, diabetes etc. High SYNTAX score is associated with increased total and cardiovascular mortality.

The aim of this study is to investigate serum heme oxygenase-1 level and SYNTAX score in patients with suspected coronary artery disease. Patients will be recruited from a single center consecutively. Blood samples will be drawn before coronary angiography. SYNTAX score will be calculated for each patient. Demographical and clinical characteristics of patients will also be recorded. Patients without coronary artery disease will be used as control group. Primary outcome measure will be to determine the relationship between HO-1 levels and SYNTAX score.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected stable coronary artery disease who are deemed to undergo coronary angiographic evaluation

Exclusion Criteria:

* Patients with history of coronary bypass or other cardiac surgery
* Patients with acute coronary syndrome
* Patients with severe comorbid illnesses including active malignancies, stage 3-5 chronic renal failure, chronic obstructive lung disease
* Patients with clinically overt infectious or inflammatory diseases
* Patients taking medications that possibly interact with heme metabolism
* patients with hemoglobinopathies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients from a single center with suspected stable coronary artery disease who are deemed to undergo coronary angiographic evaluation will be included in the study. Patients will be recruited in a non randomized fashion.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Relationship between serum heme oxygenase-1 enzyme level and SYNTAX score | 3 months
  Correlation between serum heme oxygenase levels (in pg/ml) and angiographically determined SYNTAX scores (no unit) will be determined statistically.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No